CLINICAL TRIAL: NCT00789126
Title: A Phase 1, Randomized, Double-Blind, Single-Dose Escalation Study and Multiple-Dose Escalation Study of VX-509 in Healthy Subjects
Brief Title: Single and Multiple Dose Escalation Study of VX-509 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: George Spencer-Green, MD, MS, Vertex Pharmaceuticals
Allocation: Randomized | Masking: Double
Other Study IDs: VX08-509-002
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
MeSH Terms: interventions — 2-((2-(1H-pyrrolo(2,3-b)pyridin-3-yl)pyrimidin-4-yl)amino)-2-methyl-N-(2,2,2-trifluoroethyl)butanamide

INTERVENTIONS:
Drug: VX-509

SUMMARY:
Study to evaluate the safety and tolerability of single ascending doses and multiple ascending doses of VX-509 administered to healthy male and female subjects

DETAILED DESCRIPTION:
Part A of the study will evaluate the safety and tolerability, PK, and PD of single ascending doses of VX-509.

Part B will evaluate the safety and tolerability, PK, and PD of multiple ascending doses of VX-509 administered for 14 days.

A total of 72 subjects will be enrolled: 36 subjects in Part A and 36 subjects in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking male or healthy, non-smoking, non-pregnant female
* Able to comply with study procedures
* Male subjects must agree to use 2 highly effective methods of contraception
* Female subjects must be of documented non-child-bearing potential or must agree to use 2 highly effective methods of contraception
* No clinically significant abnormal results for physical examination or clinically significant out of range laboratory results

Exclusion Criteria:

* History of any significant illness
* Illness within 5 days before Day 1
* Regular treatment with any medications
* Any type of tobacco or nicotine use
* History of drug or alcohol abuse or addiction within 2 years before Screening visit
* Positive tuberculin skin test at Screening
* Female subjects who are lactating or planning to become pregnant during the study period or within 90 days of last dose of study drug

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2008-10

PRIMARY OUTCOMES:
Safety and Tolerability as measured by adverse events (AEs) and clinically relevant changes in laboratory values, vital signs, electrocardiograms (ECGs), and physical examination variables | Specified timepoints in the protocol

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameters (Cmax, AUC, t1/2, tmax) | Specified timepoints in the protocol
Pharmacodynamics (PD)parameters of percent and actual change from baseline for a panel of JAK-dependent biomarkers | Specified timepoints in the protocol

CONTACTS AND LOCATIONS:
Overall Officials: George Spencer-Green, MD, MS, Study Director — Vertex Pharmaceuticals Incorporated
Locations (1):
- Lenexa, Kansas, United States